CLINICAL TRIAL: NCT06764160
Title: An Open-label, Single-arm, Multi-center Study to Evaluate the Efficacy, Safety, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of Eculizumab in Chinese Participants With Refractory Generalized Myasthenia Gravis (gMG)
Brief Title: Efficacy, Safety, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of Eculizumab in Chinese Adults With gMG
Acronym: ECU-MG-304
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D7411C00003; ECU-MG-304 (Other: Alexion)
Record Dates: First submitted 2024-12-11; First posted 2025-01-08 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Generalized Myasthenia Gravis (gMG); Refractory gMG
Keywords: Generalized Myasthenia Gravis (gMG); Refractory gMG; Eculizumab
MeSH Terms: conditions — Myasthenia Gravis | interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eculizumab (Experimental): Eculizumab
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab — Participants will receive Eculizumab via intravenous (IV) infusion.

SUMMARY:
This is an open-label, single-arm, multi-center study to evaluate the efficacy, safety, PK, PD, and immunogenicity of eculizumab in Chinese participants with refractory gMG. Approximately 15 participants will be enrolled in the study.

DETAILED DESCRIPTION:
This post-approval study is an open-label, single-arm, multi-center study to evaluate the efficacy, safety, PK, PD, and immunogenicity of eculizumab in Chinese participants with refractory gMG. There will be 3 periods in this study: Screening Period (up to 4 weeks), Treatment Period (26 weeks, including an Induction Phase and a Maintenance Phase), and Safety Follow-up Period (8 weeks). The overall study duration for an individual participant is estimated to be up to 38 weeks. Approximately 15 participants will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MG must be made by the following tests:

  1. Positive serologic test for anti-AChR Abs as confirmed at Screening, and
  2. One of the following:

     1. Abnormal neuromuscular transmission demonstrated by repetitive nerve stimulation, or
     2. History of positive anticholinesterase test, eg, neostigmine test, or
     3. Participant has demonstrated improvement in MG signs on oral cholinesterase inhibitors as assessed by the treating physician
* MGFA Clinical Classification Class II to IV at Screening
* MG-ADL total score must be ≥ 6 at Screening and Day 1
* Participants who have:

  1. Failed treatment with 2 or more ISTs over one year (either in combination or as monotherapy), ie, continue to have impairment ADLs (persistent weakness, experience crisis, or unable to tolerate IST) despite ISTs or,
  2. Failed at least one IST and require chronic PE or IVIg to control symptoms, ie, participants who require PE or IVIg on a regular basis for the management of muscle weakness at least 2 cycles over last 12 months

Exclusion Criteria:

* Any untreated thymic malignancy, carcinoma, or thymoma
* History of thymectomy or any other thymic surgery within 6 months prior to Screening. Participants with a history of treated thymic malignancy or carcinoma are eligible if they meet all of the following conditions:

  1. Treatment completed > 5 years prior to the Screening Visit
  2. No recurrence within the 5 years prior to the Screening Visit
  3. No radiological indication of recurrence in a computed tomography (CT) or magnetic resonance imaging (MRI) scan, including administration of intravenous (IV) contrast, performed within 6 months of first dose on Day 1
* Weakness only affecting ocular or peri-ocular muscles (MGFA Class I)
* MG crisis at Screening (MGFA Class V). However, such participants may be rescreened with Alexion approval once they are treated and medically stable, in the opinion of the Investigator
* History of N meningitidis infection or unresolved meningococcal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-12-29 (Actual); Study Completion 2025-12-29 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of eculizumab in the treatment of refractory gMG based on the improvement in the MG-ADL | from baseline at Week 26
  The mean change of Myasthenia Gravis Activities of Daily Living Profile (MG-ADL) total score from baseline at Week 26 along with 2-sided 95% CI

SECONDARY OUTCOMES:
To assess the efficacy of eculizumab in the treatment of refractory gMG by QMG | from baseline at Week 26
  The mean change of quantitative myasthenia gravis (QMG) total score from baseline at Week 26 along with 2-sided 95% CI
To assess the efficacy of eculizumab in the treatment of refractory gMG by MGC | from baseline at Week 26
  The mean change of myasthenia gravis composite (MGC) total score from baseline at Week 26 along with 2-sided 95% CI
To assess the efficacy of eculizumab in the treatment of refractory gMG by MG-QoL 15r | from baseline at Week 26
  The mean change of revised Myasthenia Gravis Quality of Life 15-Item Scale (MG-QoL 15r scale) from baseline at Week 26 along with 2-sided 95% CI
To assess the efficacy of eculizumab in the treatment of refractory gMG by MG-ADL responder status | from baseline at Week 26
  The proportion of participants who achieve the Myasthenia Gravis Activities of Daily Living Profile (MG-ADL) response at Week 26, along with the 2-sided 95% CI
To assess the efficacy of eculizumab in the treatment of refractory gMG by QMG responder analysis | from baseline at Week 26
  The proportion of participants who achieve the quantitative myasthenia gravis (QMG) response at Week 26, along with the 2-sided 95% CI
To assess the safety and tolerability of eculizumab in the treatment of refractory gMG | from baseline at Week 26
  Incidence of AEs, SAEs, and AEs leading to study intervention discontinuation (onset after first infusion)
To characterize the PK of eculizumab in participants with refractory gMG | from baseline at Week 26
  Mean serum eculizumab concentrations at all scheduled visits
To characterize the PD of eculizumab in participants with refractory gMG | from baseline at Week 26
  Mean changes in serum free complement component 5 (C5) concentrations at all scheduled visits
To characterize the immunogenicity of eculizumab in participants with refractory gMG | from baseline at Week 26
  Proportion of treatment-emergent anti-drug antibody (ADA) positive participants

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Research Site, Changchun
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Qingdao
  - Research Site, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
  Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home